CLINICAL TRIAL: NCT03946371
Title: Relation Between the Volume of Subglottic Secretion and Risk of Extubation Failure in ICU Patients
Brief Title: Relation Between the Volume of Subglottic Secretion and Risk of Extubation Failure in ICU Patients (SEGEX)
Acronym: SEGEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/429
Record Dates: First submitted 2019-04-24; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Airway Extubation; Pneumonia, Bacterial; Aspiration of Subglottic Secretions
Keywords: Sub glottic secretions; Failure Extubation; endotracheal tube
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extubation Success: Patients who do not require re-intubation, upto 48 hours after a planned extubation in the adult intensive care unit.
- Extubation failure: Patients who required re-intubation within 48 hours after a planned extubation in adult intensive care unit.

SUMMARY:
This study evaluates the relation between the volume of subglottic secretion before airway extubation and the risk of extubation failure in the ICU patient.

DETAILED DESCRIPTION:
Between 10 and 20% of patients develop extubation failure (10.7% in our ICU at 2018), which is related to an increased in-hospital death rate, infections, higher costs and longer hospital stays. Tracheal secretions, LVEF<30%, MV > 7d, Weak of cough are identified as risk factors of extubation failures but are not completely performants. Avoiding reintubation remains an important clinical goal.

The subglottic secretion drainage above the cuff of an endotracheal tube is recognized as an effective method to prevent ventilator-associated pneumonia (VAP) in critically ill patients. The subglottic secretion drainage is used in a regular way in our ICU. Volume of subglottic secretion is not analysed in the scientific literature.

Study :

The investigators hypothesize that high volume of subglottic secretion before extubation is associated with high risk of extubation failure and à high risk of pneumonia post extubation.

All planned extubations in the intensive care unit after 2 days minimal of mechanic ventilation are recorded on a designated form and standard variables charted. All data will be collected retrospectively after the extubation event.

All included patients will be assigned a unique identification number (UID) by the investigator, who will secure the patient identifiers in an encrypted electronic file. The cause of extubation failure will be recorded (as identified by the attending physician on service, who is not involved in the study).

For statistical analysis, group that fail extubation, will be compared, with the group that was an extubation success. Standard demographics (age, sex), patient disease related factors (diagnosis, duration of intubation, secretions), care factors (cuff leak test, p/f ratio prior to extubation,LVEF<30% ), and post extubation care (post extubation respiratory support, stridor, blood gas, pneumonia) along with any complication during extubation and reintubation and reasons for reintubation will be collected and compared.

As two groups are being compared, bivariate analyses utilizing Chi-square tests or univariate logistic regression for categorical variables and Student t -tests for interval variables, will be done.

Investigators will perform an interim analysis at the end of 12 months and a final analysis

ELIGIBILITY:
Inclusion Criteria:

* intubated with an orotracheal tube with a subglottic aspiration for more than 24 hours
* mechanical ventilation for more than 48 hours
* planned extubations in the intensive care

Exclusion Criteria:

* age < 18 years
* terminal extubation
* Self extubation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in intensive care intubated with an orotracheal tube with a subglottic aspiration for more than 24 hours; and receiving mechanical ventilation for more than 48 hours. Planned extubations in the intensive care
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | 48 hours
  defined as a need for reintubation within 48 h after extubation
Volume of Subglottic Secretion | 24 weeks
  Quantity (ml) of pre-extubation subglottic secretion during the duration of mechanical

SECONDARY OUTCOMES:
Weaning mechanical ventilation failure | 7 days
  Use of non-invasive ventilation ( non-invasive ventilation / High-Flow Nasal Cannula) for curative purposes within 7 days after extubation or failure extubate within 72 hours (7 days if using NIV-HFNC)
Pneumonia post extubation | 7 days
  If diagnosis retained by the doctor in charge of the patient and antibiotherapy set up for a duration of more than 5 days and occurred within 7 days post extubation
Length of stay in ICU | 22 month
  Length of stay in ICU
Mortality | 28 days
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Paillot, MD, Principal Investigator — CHU Jean Minjoz
Locations (1):
- Chu Besancon, Besançon, Doubs, France